CLINICAL TRIAL: NCT02482974
Title: Conversion From Sirolimus to Everolimus in the Maintenance Treatment of Liver Transplant Recipients: A 1-year Observational Study
Brief Title: Conversion From Sirolimus to Everolimus in the Maintenance Treatment of Liver Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ilker Turan, Assoc. Prof., Ege University
Other Study IDs: 15-3.1/53
Record Dates: First submitted 2015-06-19; First posted 2015-06-26 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Liver Transplant Recipients
Keywords: Liver transplantation; Everolimus; Sirolimus; Treatment outcome; Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to determine the safety and efficacy of conversion of sirolimus to everolimus in the maintenance treatment of LT recipients. Patients will be monitored every 12 weeks after the switch of treatment for 48 weeks. The laboratory tests including hematological, renal, hepatic, and metabolic parameters will be performed at each visit. Twenty-four-hour urine creatinine clearance and proteinuria will be determined from a 24-hour urine collection at baseline and week 48.

DETAILED DESCRIPTION:
Everolimus (EVL) and sirolimus (SRL), an antagonist of mammalian target of rapamycin, has been introduced into solid organ transplantation to either replace or reduce the dose of potentially nephrotoxic calcineurin inhibitors. Although not approved for liver transplantation (LT), SRL has still been used in several LT centers. After EVL was approved by FDA and the Ministry of Health in Turkey for use in LT recipients, SRL was converted to EVL in our institution. This study aims to determine the safety and efficacy of conversion of SRL to EVL in the maintenance treatment of LT recipients.

Patients who switch from SRL to EVL will be monitored every 12 weeks after the switch of treatment for 48 weeks.

Efficacy measure will be included any observation in terms of biopsy-proven acute/chronic rejection and graft or patient loss due to rejection.

Safety evaluations will be included discontinuation of EVL and analyses of adverse events and grading laboratory abnormalities.

Laboratory evaluations will be included hematological (CBC), renal (serum creatinine, estimated glomerular filtration rate [eGFR; Modification of Diet in Renal Disease (MDRD) and Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI)], and electrolytes), hepatic (serum transaminases, alkaline phosphatase, γ-glutamyl transferase, bilirubin, and albumin), and metabolic parameters (fasting glucose, cholesterol, and triglyceride) at each visit. Twenty-four-hour urine creatinine clearance and proteinuria will be determined from a 24-hour urine collection at baseline and week 48.

For patients who were on additional immunosuppressive treatments, those medications will also be continued.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Liver transplant recipients who switch from sirolimus to everolimus

Exclusion Criteria:

* Patients who refuse the everolimus switching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with liver transplantation who switch from sirolimus to everolimus
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with advers events, biopsy-proven acute/chronic rejection, graft loss, or death from switching time to 48 weeks post-conversion. | 48 weeks

SECONDARY OUTCOMES:
Laboratory follow-up (hematological) | At baseline and Weeks 12, 24, 36, and 48
  It will include complete blood count (hemoglobin, hematocrit, leukocyte, and platelet)
Laboratory follow-up (hepatic) | At baseline and Weeks 12, 24, 36, and 48
  It will include serum transaminases, alkaline phosphatase, γ-glutamyl transferase, bilirubin, and albumin
Laboratory follow-up (renal) | At baseline and Weeks 12, 24, 36, and 48
  It will include serum creatinine, eGFR (MDRD and CKD-EPI), and electrolytes (sodium, potassium, calcium, magnesium, and phosphate)
Laboratory follow-up (metabolic) | At baseline and Weeks 12, 24, 36, and 48
  It will include fasting glucose, cholesterol, and triglyceride.
Laboratory follow-up (24-hour urine creatinine clearance) | At baseline and Week 48
Laboratory follow-up (24-hour urine proteinuria) | At baseline and Week 48
Median dose of everolimus | 48 weeks
  The median dose of everolimus to reach the therapeutic range (3 - 8 ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Turan, M.D., Principal Investigator — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)